CLINICAL TRIAL: NCT01859637
Title: Twelve-month Study on the Immunogenicity, Safety, and Efficacy of Zarzio®/Filgrastim HEXAL® in Patients With Severe Chronic Neutropenia
Brief Title: Immunogenicity, Safety, and Efficacy of Zarzio®/Filgrastim HEXAL® in Patients With Severe Chronic Neutropenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Additional pharmacovigilance activity was considered as fulfilled by the EMA.
Sponsor: Sandoz (Industry)
Collaborators: Sandoz GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP06-401
Record Dates: First submitted 2013-05-08; First posted 2013-05-22 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Severe Chronic Neutropenia
Keywords: Filgrastim, immunogenicity, severe chronic neutropenia
MeSH Terms: conditions — Neutropenia, severe chronic | interventions — Filgrastim; pegfilgrastim; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zarzio®/Filgrastim HEXAL® (Experimental): Zarzio®/Filgrastim HEXAL® was administered according to Summary of Product Characteristics (SmPC). It was provided as solution for injection in prefilled syringes with two strengths at 300 μg/0.5 ml (30 MU) and 480 μg/0.5 ml (48 MU).
  Interventions: Biological: Filgrastim

INTERVENTIONS:
Biological: Filgrastim — Zarzio®/Filgrastim HEXAL® solution for injection was provided in prefilled syringes with two strengths at 300 μg/0.5 ml (30 MU) and 480 μg/0.5 ml (48 MU). Dosage and duration for each patient is as per the recommendations in the SmPC.
  Other Names: Zarzio®/Filgrastim HEXAL®; EP2006; rhG-CSF

SUMMARY:
Purpose of the study is to investigate the safety, immunogenicity and the efficacy of Zarzio®/Filgrastim HEXAL® under chronic administration for 12 months in patients diagnosed with severe chronic neutropenia.

DETAILED DESCRIPTION:
This was a prospective, open-label, non-comparative study. Eligible patients with Severe Chronic Neutropenia received Zarzio® for 12 months. Study visits were scheduled for screening, start of treatment with Zarzio®/Filgrastim HEXAL®, 6 weeks after start of treatment and at months 3, 6, 9 and 12.

Immunogenicity assessment: Patients were screened for anti-recombinant human granulocyte colony stimulating factor (rhG-CSF) antibodies at screening (Visit 01) and at every study visit with the exception of Visit 02 (start of treatment). The evaluation of the immune response to rhG-CSF administration was made by a three-step procedure comprising a validated binding antibody screening and confirmatory radioimmunoprecipitation assay (RIP). Samples positive for binding antibodies in the confirmatory RIP assay were evaluated for neutralizing antibodies using a validated cell-based neutralization antibody assay (NAB).

Efficacy: Complete blood counts with differential white blood cell counts were performed and absolute neutrophil count (ANC) were calculated at every study visit. For each time point the neutrophil counts are summarized by the SAF set using descriptive statistics for the ANC as well as for the changes from baseline.

Safety: Adverse events are listed for the safety population set (SAF) (term, date of AE onset, date of AE resolved, AE duration, severity grade, relationship to study drug, action taken, SAE). Additionally, the following variables were also listed: Serum human chorionic gonadotropin (hCG) pregnancy test, Physical examination, vital signs (pulse, blood pressure), weight (kg), height (cm), Laboratory (hematology, clinical chemistry, urinalysis) values

ELIGIBILITY:
Inclusion criteria:

1. Patients with established congenital, cyclic or idiopathic severe chronic neutropenia having an indication for treatment with Sandoz' filgrastim according to the SmPC of the product
2. Patients ≥ 18 years of age at the day of inclusion
3. Written informed consent of patient

Exclusion criteria:.

1. Chemotherapy-induced neutropenia
2. Neutropenia in combination with confirmed diagnosis of autoimmune disease, e.g. rheumatoid arthritis, Felty's syndrome, or systemic lupus erythematosus
3. Myelodysplastic syndrome or leukemia
4. Thrombocytopenia (platelets < 50.000/mm3) or anemia (hemoglobin < 8 g/dl) with the exception of patients with Shwachman-Diamond syndrome, glycogen storage disease 1b, or Barth's syndrome
5. Sickle cell disease
6. History of malignancy of any organ system, treated or untreated, with the exception of localized basal cell carcinoma of the skin
7. For patients with congenital severe chronic neutropenia only: Any cytogenetic aberrations in bone marrow aspirates with results not older than six months suspicious for malignant transformation.
8. Known or suspected hypersensitivity to rhG-CSF products
9. Known or suspected hypersensitivity to any of the excipients of Sandoz' filgrastim product
10. Positive result of anti-rhG-CSF antibody assessment at screening
11. Absolute and relative contraindications as specified in the SmPC of Sandoz' filgrastim
12. Drug abuse, substance abuse, or alcohol abuse
13. Use of any other investigational drug at the time of enrollment, or within 30 days or 5 half-lives prior to enrollment, whichever is longer
14. Patients unwilling and/or who are not capable of ensuring compliance with the provisions of the study protocol
15. Pregnant or breastfeeding women where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum hCG laboratory test
16. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives and intrauterine devices (IUDs)). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Nakov, MD, PhD, Study Director — Sandoz Biopharmaceutical, Hexal AG, Germany
Locations (2):
- Medizinischen Hochschule (MHH) Hannover, Hanover, Germany
- Karolinska Institut, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Since there are only six patients enrolled, all the patient data is already provided in the registry.

REFERENCES:
- [Background] Dale DC, Cottle TE, Fier CJ, Bolyard AA, Bonilla MA, Boxer LA, Cham B, Freedman MH, Kannourakis G, Kinsey SE, Davis R, Scarlata D, Schwinzer B, Zeidler C, Welte K. Severe chronic neutropenia: treatment and follow-up of patients in the Severe Chronic Neutropenia International Registry. Am J Hematol. 2003 Feb;72(2):82-93. doi: 10.1002/ajh.10255. PMID 12555210
- [Background] Palmblad J, Papadaki HA. Chronic idiopathic neutropenias and severe congenital neutropenia. Curr Opin Hematol. 2008 Jan;15(1):8-14. doi: 10.1097/MOH.0b013e3282f172d3. PMID 18043240
- [Background] Zeidler C, Welte K. Hematopoietic growth factors for the treatment of inherited cytopenias. Semin Hematol. 2007 Jul;44(3):133-7. doi: 10.1053/j.seminhematol.2007.04.003. PMID 17631177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: 05-Jul-2011, last patient in: 12-Feb-2013. 2 sites (medical school and university hospital)
Groups:
- Zarzio®/Filgrastim HEXAL® (EP2006): Open label single arm. All patients received Zarzio® subcutaneously dosed as per recommendations in Summary of Product Characteristics (SmPC).
Period: Overall Study
Arm/Group | Zarzio®/Filgrastim HEXAL® (EP2006)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to treat (ITT): All patients with at least one dose EP2006. Safety population (SAF): ITT and at least one post-baseline safety assessment. Immunogenicity population: ITT and at least one available anti-rhG-CSF antibody assessment.
  No patient was excluded of any of the populations. Results presented for SAF.
Groups:
- Zarzio®/Filgrastim HEXAL®: Open label single arm. All patients received Zarzio®/Filgrastim HEXAL® subcutaneously dosed as per recommendations in SmPC.
Arm/Group | Zarzio®/Filgrastim HEXAL®
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 45.0 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5
  Latin American | 1
Region of Enrollment [Number; unit: participants]
  Sweden | 4
  Germany | 2
Severe Chronic Neutropenia (SCN) diagnosis [Number; unit: participants]
  Congenital neutropenia | 1
  Cyclic neutropenia | 1
  Idiopathic neutropenia | 4
Granulocyte Colony Stimulating Factor (G-CSF) pretreatment [Number; unit: participants]
  Yes | 6
  No | 0
Height [Median (Full Range); unit: cm] | 165.0 [159 to 174]
Weight [Median (Full Range); unit: kg] | 67.0 [55 to 98]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Anti- Recombinant Human Granulocyte Colony Stimulating Factor (rhG-CSF) Antibodies
Description: Incidence of anti-rhG-CSF antibodies was monitored. Patients were screened for anti-rhG-CSF antibodies at screening and at each study except visit 02 (start of treatment = baseline).
  Evaluation of immune response to rhG-CSF administration was made by a three-step procedure comprising a validated binding antibody screening and confirmatory radioimmunoprecipitation assay (RIP) and a validated cell-based neutralization antibody assay (NAB).
Time Frame: screening, 3, 6, 9 and 12 months
Population: Safety population (SAF): All patients with at least one dose Zarzio®/Filgrastim HEXAL® and at least one post-baseline safety assessment. All six patients were screened for anti-rhG-CSF antibodies at all six study visits, except for one missing assessment (no sample was taken for patient 0204 at Visit 03, which was an optional visit).
Measure: Number; unit: participants
Groups:
- Zarzio®/Filgrastim HEXAL®: All patients received open-label Zarzio®/Filgrastim HEXAL®
Arm/Group | Zarzio®/Filgrastim HEXAL®
Number analyzed (Participants) | 6
participants
  Visit 1 - negative | 6
  Visit 3 - negative | 5
  Visit 4 - negative | 6
  Visit 5 - negative | 6
  Visit 6 - negative | 6
  Visit 7 - negative | 6

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Patients experiencing AEs by system organ class and preferred term (PT) and number of events. Patients with more than one AE coded to the same PT were counted once per PT
Time Frame: 12 months
Population: Safety population (SAF): all patients with at least one dose Zarzio®/Filgrastim HEXAL® and at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | Zarzio®/Filgrastim HEXAL®
Number analyzed (Participants) | 6
participants | 6

3. Secondary Outcome: Change in Absolute Neutrophile Count (ANC)
Description: To evaluate the efficacy of Zarzio®/Filgrastim HEXAL® in patients with SCN in terms of changes in absolute neutrophile count (ANC).
  Change from each visit to baseline in ANC for all patients is calculated.
Time Frame: Participants were followed for a duration of 12 months and ANC was assessed at baseline, week 6, Month 3, Month 6, Month 9 and Month 12.
Population: as for outcome 2
Measure: Median (Full Range); unit: 10^9 cells/L
Arm/Group | Zarzio®/Filgrastim HEXAL®
Number analyzed (Participants) | 6
10^9 cells/L
  ANC Visit 1 Screening to Baseline (Visit 2) | -1.252 [-10.90 to 2.84]
  ANC Visit 3 Week 6 to Baseline (Visit 2) | 6.873 [-11.20 to 16.40]
  ANC Visit 4 Month 3 to Baseline (Visit 2) | -0.198 [-11.00 to 25.50]
  ANC Visit 5 Month 6 to Baseline (Visit 2) | -0.711 [-10.80 to 12.38]
  ANC Visit 6 Month 9 to Baseline (Visit 2) | 1.506 [-9.60 to 14.70]
  ANC Visit 7 Month 12 to Baseline (Visit 2) | 1.579 [-10.80 to 18.87]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Open-label Zarzio®/Filgrastim HEXAL®: All patients received open-label Zarzio®/Filgrastim HEXAL®
Arm/Group | Open-label Zarzio®/Filgrastim HEXAL®
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Zarzio®/Filgrastim HEXAL® (N=6)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) — Patient (0101) experienced severe nephrolithiasis leading to hospitalization. No action was taken with respect to the study medication; Resolved completely 17 days after onset; Not suspected to be causally related to study medication
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Zarzio®/Filgrastim HEXAL® (N=6)
Nasopharyngitis (Infections and infestations) | 3 (5)
Genital infection fugal (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (2)
Oral herpes (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (4)
Sinusitis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tonsilitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 2 (2)
Local swelling (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an Additional Pharmacovigilance Activity (MEA005). Based on interim study data, complemented with clinical data from continued global development & extensive post-marketing experience MEA005 was considered fulfilled and the study terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days